CLINICAL TRIAL: NCT00172887
Title: Needs Assessment of Long-Term Care for Psychiatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Other Study IDs: 9461700311; DOH93-TD-M-113-013
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2005-03

CONDITIONS: Mental Disorders
Keywords: Psychiatrists
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The quantity and quality of inpatient services for persons with psychiatric illness have been enhanced in the last two decades. Following the enforcement of nationwide health insurance and the Physically and Mentally Disabled Citizens Protection Act, the financial pressure of medical care for psychiatric patients is relieved, and actions related to the protection of patients' human rights have been taken. Nonetheless, problems related to psychiatric illness are not limited to symptoms. Patients' daily functions are affected and it causes continuous pressure on the family. Currently, psychiatric care places more emphasis on inpatient services. Once the patient is discharged from the hospital, related psychiatric services are not widely available, which leads to symptom exacerbation, repeated hospital admissions, increased burden to the family, etc. A provision of continuous long-term care that meets the various needs of psychiatric patients is a critical issue in current psychiatric care.

Based on a three-phase needs assessment model, the purpose of the study is to evaluate the needs of long-term care for psychiatric patients. The first phase will identify the current status of needs from the perspectives of patients and the family, psychiatric professionals, and the system. The second phase will identify the goals of long-term care for psychiatric patients. The goals will be identified by a nominal group, composed of experts related to the field of psychiatric long-term care. The third phase will determine the objectives of long-term care services for psychiatric patients. That is to determine the proper contents of long-term care services for the patients based on the goals identified in the previous phase.

The three-phase needs assessment will be carried out in a two-year period. The results of the study will provide important information to the future planning of long-term care for psychiatric patients.

DETAILED DESCRIPTION:
First, the participants were informed about how to fill in the self-report survey questionnaire. Then the participants began to complete the questionnaire. After finishing it, the participants gave the questionnaire back to the examiner.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric patient
* Must be able to read Chinese
* Caregivers of psychiatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2005-03; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Chinyu Wu, Ph.D, Study Chair — Department of Occupational Therapy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan